CLINICAL TRIAL: NCT01929174
Title: Heart Failure and Fibrosis in Adult Congenital Heart Patients With a Single Ventricle and Prior Fontan Operation.
Brief Title: Diffuse Myocardial Fibrosis in Fontan Patients
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Craig Broberg, Associate Professor, Cardiovascular Medicine, Oregon Health and Science University
Other Study IDs: OHSUIRB00009372
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Congenital Heart Disease; Single Ventricle; Myocardial Fibrosis
Keywords: Congenital heart disease; Myocardial fibrosis; Diastolic dysfunction
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: Patients undergoing catheterization for other reasons who have a normal biventricular heart.
- Single ventricle Fontan: Patients with a single functional ventricle (excluding hypoplastic left heart syndrome) palliated with a "Fontan" type operation involving passive blood flow to the lungs.

SUMMARY:
The purpose of this protocol is to measure the relaxation of the heart in subjects with single ventricles who have undergone the surgical Fontan procedure. We will do this by measuring relaxation with MRI, echocardiography, and cardiac catheterization and compare to blood levels that measure heart scarring. We will also measure relaxation before and after boluses of intravenous (IV) fluids to see if the relaxation changes when there is more fluid in the heart. Measurements of heart relaxation will be obtained from the MRI, echocardiogram, and cardiac catheterization for each patient and compared to blood markers of heart scarring. We aim to compare all of these measurements to see if we can accurately identify heart scarring and, if present, how much it correlates with impaired heart relaxation.

ELIGIBILITY:
Inclusion criteria: adult patients (age ≥18) with a previous Fontan procedure (including all variants) referred for catheterization. This includes individuals with tricuspid atresia, double inlet left ventricle, unbalanced atrioventricular septal defect, and pulmonary atresia with intact septum. Control subjects will be selected from individuals referred to the lab for evaluation/closure of a patent foramen ovale (PFO). All subjects must be willing to participate in all portions of the study and provide written informed consent.

Exclusion criteria: contraindications to MRI such as ferromagnetic objects in the chest, claustrophobia, or contraindication to gadolinium contrast (estimated creatinine clearance < 30 ml/min/1.73m2). Fontan patients with a morphologic right ventricle (namely hypoplastic left heart after a Norwood palliation) will be excluded, because of the disproportionate risk of systolic dysfunction in the morphologic right ventricle.33 Control patients with hypertension, diabetes, coronary disease, or reduced systolic function will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a single ventricle palliated with a Fontan procedure
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Myocardial fibrosis measured by the extracellular volume fraction | 1 day of single observation
  All patients will have measurements of pressure and volume before and after IV fluid administration, as well as computation of their extracellular volume fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Broberg, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science Univ., Portland, Oregon, United States